CLINICAL TRIAL: NCT03504956
Title: Coronary Atherosclerosis T1-Weighted Characterization (CATCH)
Acronym: CATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Debiao Li, PhD, Director, Biomedical Imaging Research Institute, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 45312
Record Dates: First submitted 2018-03-19; First posted 2018-04-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Coronary Atherosclerosis
Keywords: MRI technique; High Resolution MRI Technique
MeSH Terms: conditions — Coronary Artery Disease | interventions — Magnetic Resonance Imaging; Contrast Media; gadobutrol; Adrenergic beta-Antagonists; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Other): Approximately 110 healthy male/female adult "normals" or "controls" will receive non-contrast or contrast-enhanced Cardiac MRI. Imaging may include administration of contrast and a beta blocker, based upon the focus of the study at the time of the scan, as well as the safety profile of the participant.
  Interventions: Device: Cardiac MRI; Drug: Contrast; Drug: Beta blocker
- Coronary Artery Disease (CAD) Patients (Other): 40 male/female adult outpatients who are suspected of having or have been diagnosed with coronary artery disease (CAD) will receive non-contrast or contrast-enhanced Cardiac MRI. Imaging may include administration of contrast and a beta blocker, based upon the focus of the study at the time of the scan, as well as the safety profile of the participant.
  Interventions: Device: Cardiac MRI; Drug: Contrast; Drug: Beta blocker

INTERVENTIONS:
Device: Cardiac MRI — MRI with/without administration of a contrast agent and beta-blocker based upon the stage of method development, if no contraindications are present.
  Other Names: Magnetic Resonance Imaging
Drug: Contrast — The intravenous gadolinium based contrast agent to be used in this study is Gadavist (up to 0.2 mmol/kg).
  Other Names: contrast agent; Gadavist
Drug: Beta blocker — Based upon the focus of the study at the time of the scan, a beta- blocker (metoprolol), in pill form based upon blood pressure and heart rate, may be administered to some subjects to improve the heart's ability to relax and slow the heart rate. The slower heart rate may improve image quality and lessen motion artifact.
  Other Names: Metoprolol

SUMMARY:
This study proposes to develop an MRI technique named Coronary Atherosclerosis T1-weighed Characterization (CATCH) that will improve the quality and reliability of coronary atherosclerosis evaluation, as well as simplify the scanning process and significantly shorten imaging time compared with conventional imaging methods.

DETAILED DESCRIPTION:
Approximately 110 healthy male/female adult "normals" or "controls" and 40 male/female adult outpatients who are suspected of having or have been diagnosed with coronary artery disease will be recruited. All subjects will be asked to undergo either a non-contrast MRI or a contrast-enhanced MRI of the coronary artery depending upon the focus of development at the time of their participation

It is anticipated that healthy volunteers will undergo non-contrast or contrast-enhanced MRI for evaluating the image quality associated with each acquisition module of the developed technique and motion artifact associated with motion compensation strategy. For subjects receiving contrast, a total dose of up to 0.2 mmol/kg of a gadolinium based contrast agent will be injected intravenously provided all the safety requirements are met.

Subjects undergoing a contrast-enhanced MRI will be screened using the standard clinical protocol to determine whether it is safe to administer contrast. If subjects do not qualify for contrast administration, they may be asked to have a research scan without contrast.

Research MRI results will be compared with clinical diagnostic CT and/or invasive imaging studies for patients who have been evaluated with these exams at Cedars-Sinai Medical Center..

ELIGIBILITY:
Inclusion:

* Healthy Volunteers: male or female ≥ 18 years of age with a BMI<30, with no history of cardiovascular disease
* Patients: Medically stable, male or female ≥ 18 years of age who is have not suspected of having or has been diagnosed with coronary artery disease and undergone stenting or bypass surgery

Exclusion:

* Contraindications to MR imaging including mechanically, magnetically, or electrically activated implants, ferromagnetic implants and ferromagnetic foreign bodies, pregnancy.
* Inability to tolerate MR imaging secondary to an inability to hold breath for a short time or have claustrophobia.
* Non-compliant with visit instructions, including following procedure instructions
* Severe allergy to animal dander or animal-instigated asthma
* Specific to gadolinium-based contrast agents: Renal function test does not meet CSMC standard of care MRI contrast protocol requirements (GFR <45ml/min) or previous allergic reaction to gadolinium-based contrast agents.*
* Volunteers who have had four or more prior previous gadolinium contrast scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plaque to Myocardial Ratio (PMR). | Day 1
  PMR is defined as the ratio between the maximal signal intensity from a vessel wall region and the average signal from an adjacent myocardial area. Such metric is used to classify hyper-intense plaques, also known as "hot spots", which has PMR over 1.0.

SECONDARY OUTCOMES:
Stenosis level (patient group only) | Day 1
  Stenosis level will be evaluated at the vascular segments with visible lumen narrowing in each patient. The extent of a stenosis will be measured and recorded as a percentage, ranging from 0% to 100%, with 100% representing a complete occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Debiao Li, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No